CLINICAL TRIAL: NCT06492967
Title: Latin American Lifestyle Intervention Initiative to Reduce the Risk and Prevent Cognitive Impairment.
Brief Title: LatAm-FINGERS Initiative for Cognitive Change
Acronym: LatAmFINGERS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la Lucha contra las Enfermedades Neurológicas de la Infancia (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Prof. Ricardo F. Allegri, MD., PhD., PhD, Fundación para la Lucha contra las Enfermedades Neurológicas de la Infancia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SG-21-715176-LatAm-FINGERS
Record Dates: First submitted 2023-05-30; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; Brain Diseases; Lifestyle
MeSH Terms: conditions — Alzheimer Disease; Brain Diseases

STUDY DESIGN:
Intervention Model Description: Multicenter study with blind evaluators, evaluating the feasibility of a lifestyle intervention over two years.
Who Masked: Outcomes Assessor
Masking Description: Multicenter study with blind evaluators, evaluating the feasibility of a lifestyle intervention over two years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systematic Lifestyle Intervention (Experimental): Lifestyle modification program that involves participants completing structured activities that target diet, physical exercise, and intellectual and social stimulation.
  Interventions: Behavioral: Systematic Lifestyle Intervention
- Flexible Lifestyle Intervention (Experimental): Lifestyle modification program that is developed by the participant to meet his/her specific needs.
  Interventions: Behavioral: Flexible Lifestyle Intervention

INTERVENTIONS:
Behavioral: Systematic Lifestyle Intervention — Lifestyle intervention that involves providing participants with education, support, and tangible tools to assist them in developing and carrying out healthier lifestyle practices.
  Other Names: Systematic Lifestyle Intervention (SLI)
  Arms: Systematic Lifestyle Intervention
Behavioral: Flexible Lifestyle Intervention — Lifestyle intervention that involves a structured program of diet, physical and cognitive exercise, and management of cardiometabolic risks.
  Other Names: Flexible Lifestyle Intervention (FLI)
  Arms: Flexible Lifestyle Intervention

SUMMARY:
Currently, 40% of global dementia cases can be prevented through lifestyle changes, with Latin America having a 56% potential reduction due to its high-risk factors. At the moment, there are no medications that halt the clinical expression of dementia.

LatAm-FINGERS, a multicenter study across 12 Latin American countries, aims to study the feasibility of an intervention modifying lifestyle in individuals aged 60 to 77 at risk of dementia. Success could influence public policy on clinical care for older adults.

DETAILED DESCRIPTION:
Today we know that 40% of dementia cases worldwide can be prevented through lifestyle modification. If we look at Latin America, this number is 56%. Latin America is a region with high-risk factors for dementia due to weakened socioeconomic infrastructure, an impoverished healthcare system, and low average education levels in the region. Additionally, we know that cardiovascular health is an important factor in the development of dementia.

Under this scenario, LatAm-FINGERS is a multicenter study designed to prevent memory decline through lifestyle modification in people aged 60 to 77 at risk of dementia. Twelve Latin American countries are participating (Argentina, Bolivia, Brazil, Chile, Colombia, Dominican Republic, Mexico, Puerto Rico, Uruguay, Costa Rica, Ecuador, and Peru), with 100 individuals per center. These individuals are randomly assigned to two groups: (1) a group making systematic lifestyle changes (physical and cognitive training, implementation of the Mediterranean-dietary approach to stop hypertension (DASH) Intervention for Neurodegenerative Delay (MIND) diet, socialization, and regular health check-ups) and (2) a group receiving regular health advice.

The main objective of LatAm-FINGERS is to determine if this intervention is feasible in Latin America. Secondarily, we want to test if this lifestyle change can lead to improvements in participants' cognition over time (2 years).

If successful, the results of this study will have large-scale implications for public policy regarding the standard of clinical care and prescriptive practices for a fast-growing and vulnerable population of older adults.

LatAm-FINGERS is based on the Finnish Geriatric Intervention Study to Prevent Cognitive Impairment and Disability (FINGER), which demonstrated that lifestyle modification promotes positive changes in memory and attention. Additionally, our study is aligned with the U.S. Study to Protect Brain Health Through Lifestyle Intervention to Reduce Risk (U.S. POINTER), which is conducting a similar intervention in the United States.

This project is fully funded by the Alzheimer's Association.

ELIGIBILITY:
Inclusion Criteria

* Age: 60-77 years.
* Cardiovascular Risk Factors, Aging, and Incidence of Dementia (CAIDE) Risk Score > 6.
* Mini-Mental State Examination (MMSE) z score between 0 and -1.5 OR
* CERAD Word List Learning Task (10 word x 3 repetitions) < 0 z score OR
* CERAD (delayed word list recall) < z score < 0

Exclusion Criteria

* MMSE < 20
* Dementia
* Any medical condition that affects the participant's safety.
* Severe osteoarticular problems that preclude the implementation of the physical activity intervention outlined in the protocol, such as, for example: osteoarthrosis of the knee(s), coxofemoral, or other.
* Significant neurological disease, including dementia, cognitive impairment, Parkinson's disease, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis or history of significant head injury with persistent neurological sequelae or structural brain abnormalities, major depressive disorder within the last 2 months, history of bipolar disorder or schizophrenia according to Diagnostic and Statistical Manual of Mental Disorders V (DSM V) criteria.
* Severe cardiovascular disease, including heart failure, clinically significant aortic stenosis, history of uncontrolled acute myocardial infarction (AMI) or angina and Cardiac rhythm disorders: g3 conduction block, uncontrolled arrhythmia, alterations in Q wave, S waver and T wave segment or QT segment and auricular fibrillation (AF) of less than one year of evolution, venous thrombosis or pulmonary thromboembolism (PTE) of less than 6 months of evolution and any pathology that in clinical judgment compromises the intervention of physical activity.
* Body Mass Index >40
* Cerebral vascular disease in the last 2 years.
* Insulin-dependent diabetes mellitus.
* Pulmonary disease requiring oxygen and/or steroids.
* Renal disease defined as increased renal glomerular filtration rate <60ml/min/1.73mt2 or albumin excretion rate (AER) > 30mg/24 hrs.
* Clinically significant laboratory abnormalities as judged by the investigator.
* History within the last 2 years of treatment for primary or recurrent malignant disease.
* History of hip fracture, knee replacement, or spinal surgery within the last 6 months.
* Being in cardiopulmonary rehabilitation.
* History of bariatric surgery.
* Cardiac surgery in the last year.
* Severe sensory loss or loss of communication skills.
* No schooling.
* Use of psychoactive medications within the past 3 months, including tricyclic antidepressants, antipsychotics, psychotropic mood-stabilizing agents (e.g., lithium salts), psychostimulants, opioid analgesics, antiparkinsonian medications, anticonvulsant medications (except gabapentin and pregabalin for non-convulsant indications), systemic corticosteroids, or medications with significant central anticholinergic activity; in the absence of major depression, stable doses of selective serotonin reuptake inhibitors or serotonin and norepinephrine reuptake inhibitors are permitted.
* Active participation in another intervention study.
* History of alcoholism or substance abuse in the last 2 years, according to DSM V criteria.

Ages: 60 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Reach | Up to 2 years
  It refers to the effectiveness of recruiting the target population. It will be measured by the ratio of randomized participants versus the ratio of screen-failures.
Implementation | Up to 2 years
  Adherence rate of participants to the protocol in both arms. It will be measured through the percentage of attendance to group meetings, attendance to physical and cognitive training sessions, and completion of dietary records.
Maintenance | Up to 2 years
  It consists of each center's ability to sustain the intervention. It will be measured through the percentage of subjects who complete outcome measures at each trial event (baseline, 6, 12, 18, and 24 months).

SECONDARY OUTCOMES:
Global cognition | Up to 2 years
  Global cognitive function will be obtained from a composite score derived from subtest scores on the LatAm Neuropsychological Test Battery (LatAm-NTB) that includes: Free and Cued Selective Reminding Test, Logical Memory, Digit Span, Concept Shifting Test, Digit Symbol Substitution Test, Semantic and phonological fluency, Trial Making Test, Stroop Test.
  Scores from each individual test will be converted to z-scores that typically range from -3 to 3, with higher scores reflecting better performance, and averaged to form a composite.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Francisco Allegri, MD, Ph.D, Principal Investigator — Fleni Neurological Institute, Buenos Aires, Argentina; Lucía Crivelli, Ph.D, Principal Investigator — Fleni Neurological Institute, Buenos Aires, Argentina; Gustavo Emilio Sevlever, MD, Ph.D, Principal Investigator — Fleni Neurological Institute, Buenos Aires, Argentina; María Isabel Cusicanqui, MD, Principal Investigator — Centro Neurológico Mente Activa, La Paz, Bolivia; Ricardo Nitrini, MD, Ph.D, Principal Investigator — University of São Paulo School of Medicine, São Paulo, Brazil; Paulo Caramelli, MD, Ph.D, Principal Investigator — Universidade Federal de Minas Gerais, Belo Horizonte, Brazil; Carolina Delgado Derio, MD, MSc, Principal Investigator — Hospital Clínico Universidad de Chile, Santiago, Chile; Francisco Lopera, MD, Ph.D, Principal Investigator — Antioquia University, Colombia; Jorge Mario Leon-Salas, MD, Principal Investigator — GBHI, TCD. Hospital Clínica Bíblica, San José, Costa Rica; Lissette Duque-Peñailillo, MD, Principal Investigator — Neuromedicenter, Quito, Ecuador; Ana Luisa Sosa, MD, Ph.D, Principal Investigator — Instituto Nacional de Neurología y Neurocirugía Manuel Velasco Suárez, México; Nilton Custodio, MD, Ph.D, Principal Investigator — Instituto Peruano de Neurociencias, Lima, Perú; Ivonne Z. Jiménez-Velázquez, MD, Principal Investigator — Universidad de Puerto Rico, San Juan, Puerto Rico; Daisy Acosta, MD, Ph.D, Principal Investigator — Universidad Nacional Pedro Henriquez Urena (UNPHU), Santo Domingo, Dominican Republic; Ana María Charamelo Baietti, Ph.D, Principal Investigator — Facultad de Medicina-Hospital de Clínicas, Universidad de la República, Montevideo, Uruguay; Ricardo Francisco Allegri, MD, Ph.D, Study Chair — Fleni Neurological Institute, Buenos Aires, Argentina; Paulo Caramelli, MD, Ph.D, Study Chair — Universidade Federal de Minas Gerais, Belo Horizonte, Brazil; Francisco Lopera, MD, Ph.D, Study Chair — Antioquia University, Colombia; Ricardo Nitrini, MD, Ph.D, Study Chair — University of São Paulo School of Medicine, São Paulo, Brazil; Gustavo Emilio Sevlever, MD, Ph.D, Study Chair — Fleni Neurological Institute, Buenos Aires, Argentina; Ana Luisa Sosa, MD, Ph.D, Study Chair — Instituto Nacional de Neurología y Neurocirugía Manuel Velasco Suárez, México; Ismael Calandri, MD, Study Chair — Fleni Neurological Institute, Buenos Aires, Argentina; Rosa María Salinas, MD, Ph.D, Study Chair — Instituto Nacional de Neurología y Neurocirugía Manuel Velasco Suárez, México; Claudia Suemoto, MD, Ph.D, Study Chair — University of São Paulo Medical School, São Paulo, Brazil; Lina Marcela Velilla, Ph.D, Study Chair — Antioquia University, Colombia; Mônica Sanches Yassuda, Ph.D, Study Chair — University of São Paulo School of Medicine, São Paulo, Brazil; Lucía Crivelli, Ph.D, Study Chair — Fleni Neurological Institute, Buenos Aires, Argentina; Sonia Maria Dozzi Bruki, MD, Ph.D, Study Chair — University of São Paulo School of Medicine, São Paulo, Brazil
Locations (13):
- Fleni, Ciudad Autonoma de Buenos Aire, Argentina
- Centro Neurológico Mente Activa, La Paz, Bolivia
- Brazil (2):
  - Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - University of Sao Paulo School of Medicine, São Paulo
- Hospital Clínico Universidad de Chile, Santiago, Chile
- Antioquia University, Antioquia, Colombia
- Hospital Clínica Bíblica, San José, Costa Rica
- Universidad Nacional Pedro Henriquez Urena (UNPHU), Santo Domingo, Dominican Republic
- Neuromedicenter - Cognitive Disorders Unit, Quito, Ecuador
- Instituto Nacional de Neurología y Neurocirugía Manuel Velasco Suárez, Mexico City, Mexico
- Instituto Peruano de Neurociencas, Lima, Peru
- Universidad de Puerto Rico, San Juan, Puerto Rico
- Clínica de la Memoria - Hospital Británico, Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crivelli L, Calandri IL, Suemoto CK, Salinas RM, Velilla LM, Yassuda MS, Caramelli P, Lopera F, Nitrini R, Sevlever GE, Sosa AL, Acosta D, Baietti AMC, Cusicanqui MI, Custodio N, De Simone SD, Derio CD, Duque-Penailillo L, Duran JC, Jimenez-Velazquez IZ, Leon-Salas JM, Bergamo Y, Clarens MF, Damian A, Demey I, Helou MB, Marquez C, Martin ME, Martin MDGM, Querze D, Surace EI, Acosta-Egea S, Aguirre-Salvador E, de Souza LC, Cancado GHDCP, Brucki SMD, Friedlaender CV, Gomes KB, Gutierrez M, Rios CL, Galindo JGM, Montesinos R, Nunez-Herrera A, Ospina-Henao S, Rodriguez G, Masson VR, Sanchez M, Schenk CE, Soto L, Barbosa MT, Tosatti JAG, Vicuna Y, Espeland M, Hakansson K, Kivipelto M, Baker L, Snyder H, Carrillo M, Allegri RF. Latin American Initiative for Lifestyle Intervention to Prevent Cognitive Decline (LatAm-FINGERS): Study design and harmonization. Alzheimers Dement. 2023 Sep;19(9):4046-4060. doi: 10.1002/alz.13101. Epub 2023 May 19. PMID 37204054
- See also: Project summary. — https://www.fleni.org.ar/fingers/